CLINICAL TRIAL: NCT04474990
Title: VP-VLY-686-3303: Single-Patient Expanded Access Protocol for Tradipitant In A Single Patient With Gastroparesis
Brief Title: Single-Patient Expanded Access Protocol for Tradipitant In A Single Patient With Gastroparesis
Status: Available | Type: Expanded Access
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VP-VLY-686-3303
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Gastroparesis; Diabetic Gastroparesis
Keywords: gastroparesis; idiopathic; diabetic; tradipitant; nausea; vomiting; stomach; motility; functional; NK-1 antagonist; neurokinin 1 receptor; substance p; expanded access
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Tradipitant — NK-1 Receptor antagonist

SUMMARY:
Primary Objective: To treat a single patient with gastroparesis who has requested expanded access with tradipitant

DETAILED DESCRIPTION:
This is a single-patient extended access treatment protocol to be conducted in the United States. Investigator-Physician has determined patient satisfies expanded access inclusion criteria and has requested expanded access to tradipitant.

Patient will be given open label tradipitant 85 mg to be taken twice daily at 12 hour intervals for long term treatment. Patient can fill out daily web-based symptom diaries on a voluntary basis and report any adverse events to Investigator-Physician.

Primary Objective:

-To treat a single patient with gastroparesis who has requested expanded access with tradipitant

Secondary Objectives:

* To monitor the efficacy of tradipitant in reducing individual symptoms associated with gastroparesis in this single patient
* To monitor the safety of tradipitant in a patient with gastroparesis by assessing adverse events in this single patient

ELIGIBILITY:
Inclusion Criteria:

* Identified subject who requested expanded access
* Diagnosed with gastroparesis
* Demonstrated delayed gastric emptying
* Presence of moderate to severe nausea
* Patient does not qualify for or does not have access to other clinical trials with tradipitant;

Exclusion Criteria:

* Another active disorder or treatment which could explain or contribute to symptoms of gastroparesis
* A positive test for drugs of abuse at the screening or evaluation visits;
* Exposure to any investigational medication in the past 60 days other than tradipitant
* Gastrectomy, fundoplication, vagotomy, pyloroplasty, bariatric surgery, or gastric stimulation device surgically implanted within the last year
* Any other reason as determined by the Investigator which may lead to an unfavorable risk-benefit ratio to treatment;

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Vanda Investigational Site, Maitland, Florida
  - Vanda Investigational Site, Tampa, Florida
  - Vanda Investigational Site, Wauconda, Illinois
  - Vanda Investigational Site, Wichita, Kansas
  - Vanda Investigational Site, Louisville, Kentucky
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, Chesterfield, Missouri
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, Tulsa, Oklahoma
  - Vanda Investigational Site, Philadelphia, Pennsylvania
  - Vanda Investigational Site, Nashville, Tennessee
  - Vanda Investigational Site, Houston, Texas
  - Vanda Investigational Site, Plano, Texas
  - Vanda Investigational Site, Spokane, Washington